CLINICAL TRIAL: NCT02705430
Title: Effect of EPA-DHA Supplementation, Life Style Modification or Standard Treatment on Clinical Outcome and Lipid Membrane Composition in Type 2 Diabetic Patients: a 3 Months Perspective Randomized Pilot Study.
Brief Title: Effect of EPA-DHA Supplement, Life Style Modification Standard Treatment on Clinical Outcome Lipid Membrane Composition in Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Pierre Singer, Professor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0248-15-RMC
Record Dates: First submitted 2016-03-06; First posted 2016-03-10 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (No Intervention): Group A will continue their actual therapy (control).
- B (Experimental): Group B will continue their standard therapy with additional stress management application only using a mobile phone (Eco Fusion Mentally) for 3 months of the study
  Interventions: Behavioral: Stress management phone application (Eco Fusion Mentally); Device: mobile phone
- C (Experimental): Group C will continue their standard therapy with additional life style program using a mobile phone (Eco Mentally and NewMe) for 3 months of the study
  Interventions: Behavioral: life style program using a mobile phone (Eco Mentally and NewMe); Device: mobile phone
- D (Experimental): Group D will continue their standard therapy plus additional life style program using a mobile phone with additional supplemental EPA and DHA capsules of 2 g/day to be taken daily for the 3 months of the study
  Interventions: Dietary Supplement: EPA and DHA capsules of 2 g/day; Behavioral: life style program using a mobile phone (Eco Mentally and NewMe); Device: mobile phone

INTERVENTIONS:
Dietary Supplement: EPA and DHA capsules of 2 g/day — EPA and DHA capsules of 2 g/day
  Arms: D
Behavioral: Stress management phone application (Eco Fusion Mentally) — Stress management phone application (Eco Fusion Mentally)
  Arms: B
Behavioral: life style program using a mobile phone (Eco Mentally and NewMe) — life style program using a mobile phone (Eco Mentally and NewMe)
  Arms: C; D
Device: mobile phone — mobile phone
  Arms: B; C; D

SUMMARY:
The aim of the present study is: to examine some of the mechanisms by which a change in life style alone or supplemented with a diet supplemented in n-3 PUFA, and associated with this computerized life style regulation reduces the development of diabetic complication in a small population based study.

(The NewMe™ / Eco-fusion, Ltd is a science-driven lifestyle change program for better living -www.eco-fusion.com)

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 18-80 years of age.
2. Have been diagnosed with type 2 diabetes more than nine months before study entry, and, despite having been given standard dietary advice by dietitian, doctor, or nurse and prescribed oral hypoglycaemic agents, insulin, or both.
3. Have persistent unsatisfactory glycaemic control defined as HbA1c more than 7%.
4. Participants should have at least two of the following three characteristics:

   1. Overweight or obesity (body mass index ≥25),
   2. Hypertension (currently prescribed antihypertensive drugs or blood pressure >140/90 mm Hg despite optimized antihypertensive drug treatment),
   3. Dyslipidaemia (currently prescribed lipid modifying drugs) or one or more of:

   <!-- -->

   1. total cholesterol >5.2 mmol/l,
   2. low density lipoprotein cholesterol >3.5 mmol/l,
   3. triglycerides >2.0 mmol/l,
   4. high density lipoprotein cholesterol <1.0 mmol/l (despite optimised lipid modifying drug treatment).

Exclusion Criteria:

1. Pregnancy
2. Serious chronic illness.e.g cancer
3. End stage renal failure
4. Amputation
5. Stroke
6. Severe retinal microangiopathy
7. Pancreas transplantation
8. HbA1c <7%
9. Requires diet only treatment
10. They are too busy with work

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c < 7% | 3 months
  To attain individualized HbA1c < 7% goal

SECONDARY OUTCOMES:
Changes in hypoglycaemic drugs (type and dose), | 3 months
Blood pressure< 140\80 mmHg | 3 months
Fasting plasma glucose | 3 months
lipid profile. LDL cholesterol ,100 mg/dL; triglycerides ,150 mg/dL; HDL cholesterol .40 mg/dL for men; HDL cholesterol .50 mg/dL for women. | 3 months
Lipid membrane fatty acid composition analysis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Singer, Professor, Principal Investigator — Head of General Intensive care unit
Locations (1):
- Rabin medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No